CLINICAL TRIAL: NCT03834805
Title: Monitoring of Fetal Lung Elasticity by Elastography Between 24 and 39 Weeks
Acronym: ELASTOPULM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: API/2018/95
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2020-05

CONDITIONS: Pregnant Woman

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women with a normal pregnancy (Experimental): Assesment of fetal lung and liver stiffness with 2D Ultrasounds Shear Wave Elastography
  Interventions: Other: lung and liver elastography measurement of fetus

INTERVENTIONS:
Other: lung and liver elastography measurement of fetus — Other: lung and liver elastography measurement of fetus

SUMMARY:
The objective of the study is to evaluated the evolution of the LLE ratio (Lung to Liver Elastography ratio) during normal pregnancy

ELIGIBILITY:
Inclusion Criteria:

* major pregnant women
* singleton pregnancy

Exclusion Criteria:

foetus:

* fetal pulmonary disease
* fetal liver disease
* chromosome fetal abnormalities
* fetal growth restriction

mother:

* BMI>30 in beginning of pregnancy
* premature ruptured membranes
* high blood pressure
* pre-eclampsia
* gestational diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 74 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Change of Lung to liver Elastography ratio (LLE ratio) between 24 and 39 weeks of amenorrhea | measurements at: 24, 28, 32, 36, 39 weeks of amenorrhea (WA)
  Evolution of the fetal lung elasticity coefficient measured in kilopascals (kPa) compared to the fetal liver elasticity

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Jean Minjoz, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nallet C, Pazart L, Cochet C, Vidal C, Metz JP, Jacquet E, Gorincour G, Mottet N. Prenatal quantification of human foetal lung and liver elasticities between 24 and 39 weeks of gestation using 2D shear wave elastography. Eur Radiol. 2022 Aug;32(8):5559-5567. doi: 10.1007/s00330-022-08654-1. Epub 2022 Mar 10. PMID 35267093